CLINICAL TRIAL: NCT06569056
Title: A Multi-center, Randomized, Double-blind, Active Controlled, Parallel Groups, Phase III Study to Evaluate the Efficacy and Safety of HRS-8427 in the Treatment of Adults With Complicated Urinary Tract Infection, Including Acute Pyelonephritis
Brief Title: A Trial of HRS-8427 in the Treatment of Adults With Complicated Urinary Tract Infection, Including Acute Pyelonephritis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HRS-8427-302
Record Dates: First submitted 2024-08-22; First posted 2024-08-23 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2024-10

CONDITIONS: Complicated Urinary Tract Infection(cUTI), Including Acute Pyelonephritis(AP)
MeSH Terms: interventions — Cilastatin, Imipenem Drug Combination; Imipenem

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HRS-8427; Imipenem and Cilastatin Sodium placebo (Experimental)
  Interventions: Drug: HRS-8427; Drug: Imipenem and Cilastatin Sodium placebo
- Imipenem and Cilastatin Sodium; HRS-8427 placebo (Active Comparator)
  Interventions: Drug: Imipenem and Cilastatin Sodium; Drug: HRS-8427 placebo

INTERVENTIONS:
Drug: HRS-8427 — Dosing frequency: for 7-14 days; dose adjustments of subjects with reduced function include reduced doses
  Arms: HRS-8427; Imipenem and Cilastatin Sodium placebo
Drug: Imipenem and Cilastatin Sodium — Dosing frequency: for 7-14 days; dose adjustments of subjects with reduced function include reduced doses
  Arms: Imipenem and Cilastatin Sodium; HRS-8427 placebo
Drug: HRS-8427 placebo — Dosing frequency: for 7-14 days; dose adjustments of subjects with reduced function include reduced doses
  Arms: Imipenem and Cilastatin Sodium; HRS-8427 placebo
Drug: Imipenem and Cilastatin Sodium placebo — Dosing frequency: for 7-14 days; dose adjustments of subjects with reduced function include reduced doses
  Arms: HRS-8427; Imipenem and Cilastatin Sodium placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of HRS-8427 in patients with complicated urinary tract infection, including acute pyelonephritis.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide a written informed consent before the study, fully understand the study and be able to complete the study according to the protocol;
2. Male and female, ≥18 years;
3. Judged by the investigator, clinical diagnosis with cUTI or AP, expectation that the patients will require hospitalization and initial treatment with intravenous antibiotics;
4. Urine specimen with evidence of pyuria；
5. Have urine culture specimen obtained within 48 hours prior to randomization;
6. 48 hours before random, allowing a short course of antimicrobial drug treatment is less than 24 hours (random rate ≤25%)
7. Women of childbearing potential must have a negative serum pregnancy test before first dose, must be non-lactating. Fertile female subjects or male subjects whose partner is a fertile female agree to use highly effective form of contraception, with no plan of birth, sperm/ovum donation from the time of signed ICF till 14 days after end of treatment.

Exclusion Criteria:

1. History of significant hypersensitivity or allergic reaction to any β-lactam, or any β-lactamase inhibitors;
2. Known history of immune deficiency disease or receive immunocompromising treatment;
3. Severe cardiovascular and cerebrovascular diseases with clinical significance and unstable condition or uncontrolled;
4. Known or suspected central nervous system disorder or other factors that may predispose to seizures or lower the seizures onset threshold;
5. Presence of any known or suspected disease or condition that, in the opinion of the Investigator, may confound the assessment of efficacy;
6. Uncomplicated lower urinary tract infection;
7. Suspected or confirmed urinary tract symptoms caused by acute/chronic prostatitis, orchitis, epididymitis or sexually transmitted diseases as determined by medical history and/or physical examination;
8. Patients received cancer treatment within 4 weeks before randomization or planned treatment during the study period;
9. Systemic antimicrobial therapy other than the investigational drug need to be used during the study period, with the exception of topical or single oral dose of antifungal treatment
10. Urinary tract surgery prior to 7 days before randomization or surgery planned during the study period;
11. Indwelling catheter or urinary apparatus, the researchers determine drug treatment period cannot be removed;
12. Receipt of potentially effective systemic antibacterial therapy for a continuous duration of ≥24 hours during the previous 48 hours prior to the randomization;
13. History of pelvis or urinary tract trauma prior to the randomization;
14. Patients had severe trauma or received major surgery prior to the randomization;
15. Impairment of renal function with estimated glomerular filtration rate or Creatinine Clearance <15 mL/min ;
16. Laboratory abnormalities in baseline specimens obtained at screening;
17. A QTcF interval prolongation at screening or abnormalities with clinical significance and may cause obvious safety risk to the subjects;
18. Known urine culture with at least one Gram-Negative uropathogen at ≥105 colony-forming units(CFU)/mL unsusceptible to Imipenem and Cilastatin Sodium, or only identify Gram-positive uropathogen, or confirmed fungal urinary tract infection with ≥103CFU/mL;
19. Likely to require the use of antibiotic drug prevention after treatment;
20. Suspected of sepsis, producing life-threatening organ dysfunction;
21. Estimated survival within 6 weeks or rapidly progressive or end stage disease with high mortality rate;
22. Drug abuse prior to the randomization;
23. Participated in a previous clinical study related to HRS-8427 and used HRS-8427 or have participated in another clinical study within 4 weeks before randomization and used a study drug containing the active ingredient;
24. Judgment of the Investigator, other reasons unsuitable for study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 578 (Estimated)
Dates: Start 2024-09-25 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants With Composite Response of Microbiological Eradication and Clinical Response at Test of Cure (TOC) | Test of cure (TOC; 7 days after end of treatment [EOT], equivalent to Study Day 14 to 21)

SECONDARY OUTCOMES:
Percentage of Participants With Composite Response of Microbiological Eradication and Clinical Response at Early Assessment（EA）、End of Treatment（EOT）and Late Follow-Up (LFU) | EA : Day 4、EOT: Day 7 to Day 14、LFU：Day 21 to Day 28
Percentage of Participants With Microbiological Eradication at EA 、EOT、TOC and LFU | EA : Day 4、EOT: Day 7 to Day 14、TOC:Day 14 to Day 21、LFU：Day 21 to Day 28
Percentage of Participants With Microbiological Eradication at EA 、EOT、TOC and LFU Per Uropathogen | EA : Day 4、EOT: Day 7 to Day 14、TOC:Day 14 to Day 21、LFU：Day 21 to Day 28
Percentage of Participants With Clinical Response at EA 、EOT、TOC and LFU | EA : Day 4、EOT: Day 7 to Day 14、TOC:Day 14 to Day 21、LFU：Day 21 to Day 28
Percentage of Participants With Clinical Response at EA 、EOT、TOC and LFU Per Uropathogen | EA : Day 4、EOT: Day 7 to Day 14、TOC:Day 14 to Day 21、LFU：Day 21 to Day 28
Number of Participants With Adverse Events | Day 21 to Day 28

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Huashan Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided